CLINICAL TRIAL: NCT03530280
Title: Effect of Pregabalin or Adductor Canal Block on Postoperative Analgesia After Arthroscopic Anterior Cruciate Ligament Reconstruction (ACL)
Brief Title: Effect of Pregabalin or Adductor Canal Block on Postoperative Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Diskapi Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Fatma Kavak Akelma, specialist doctor, Ankara Diskapi Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: pregabalin
Record Dates: First submitted 2018-03-26; First posted 2018-05-21 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Postoperative Pain After Knee Arthroscopy
Keywords: pregabalin; adductor canal block; postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- pregabalin (lyrica) (Active Comparator): pregabalin (lyrica) 150 mg preoperative 1 hour before and the postoperative sham block will perform.
  Interventions: Drug: pregabalin (lyrica)
- placebo group (Placebo Comparator): a placebo capsule 1 hour before surgery and the postoperative sham block will perform.
  Interventions: Drug: Placebo oral tablet
- adductor channel block group (Active Comparator): A preoperative placebo capsule will be given.This group will receive postoperative adductor channel block including 10 mL of 0.25% bupivacaine with 5 μg/mL epinephrine
  Interventions: Drug: adductor canal block including bupivacaine

INTERVENTIONS:
Drug: pregabalin (lyrica) — preoperative pregabalin and the postoperative sham block will perform.
  Arms: pregabalin (lyrica)
Drug: Placebo oral tablet — The preoperative placebo oral tablet and the postoperative sham block will perform.
  Arms: placebo group
Drug: adductor canal block including bupivacaine — The preoperative placebo oral tablet and adductor channel block including 10 mL of 0.25% bupivacaine with 5 μg/mL epinephrine
  Arms: adductor channel block group

SUMMARY:
arthroscopically Anterior Cruciate Ligament Reconstruction (ACL) under spinal anesthesia were included in this study.

DETAILED DESCRIPTION:
Patients who American Society of Anesthesiologists (ASA) classification I to II scheduled to undergo arthroscopically assisted ACL reconstructions under spinal anesthesia are included in this study. The first group is administered 150 mg oral pregabalin 1 hour before surgery and the postoperative sham block was performed with an ultrasound probe. The second group is the control group; patients in this group are administered a placebo capsule 1 hour before surgery and sham block was performed with an ultrasound probe.The third group is administered a placebo capsule 1 hour before surgery and postoperative adductor canal block is performed. All patients will be received postoperative a tramadol i.v. patient control analgesia device. At the end of 24 hours, the total amount of tramadol consumed by the patient will be recorded from the patient control analgesia. NRS score, white fast track, satisfaction will be questioned.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 and 70 years
* American Society of Anesthesiologists I or II
* Scheduled to undergo knee arthroscopy

Exclusion Criteria:

* allergic to any medicines
* History of drug or alcohol abuse,
* Opioids or sedative medications
* History of psychiatric conditions
* Pregnant or lactating women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
11-point numerical rating scale (NRS) | 24 hours
  11-point numerical rating scale for pain (0='no pain' and 10='worst pain possible pain') were explained.
tramadol consumption | 24 hours
  24 hours tramadol consumption will be recorded as milligrams

CONTACTS AND LOCATIONS:
Locations (1):
- Diskapi Teaching and Research Hospital, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No